CLINICAL TRIAL: NCT02900157
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of MEDI9090 in Subjects With Advanced Solid Tumors
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of MEDI9090 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00055
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumor; Immunotherapy; MEDI9090; MEDI4736; Durvalumab
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEDI9090 (Experimental)
  Interventions: Biological: MEDI9090; Biological: Durvalumab

INTERVENTIONS:
Biological: MEDI9090 — MEDI9090 will be administered by IV infusion
Biological: Durvalumab — Durvalumab as a single agent will be administered by IV infusion after patients have completed the prescribed doses of Medi9090.

SUMMARY:
This is an open-label, study of MEDI9090 to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of MEDI9090 in adult subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* 18 years and older
* Must have histologic documentation of advanced solid tumors
* Must have received and have progressed, are refractory or, intolerant to standard therapy and must not have a curative therapy option

Exclusion Criteria:

* Concurrent enrollment in another clinical study
* Prior participation in clinical studies that include durvalumab alone or in combination
* Concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting infusion related reactions | First dose of study medication through 30 days after the first dose of study medication
Number of subjects that develop changes in detectable antidrug antibodies to MEDI9090 | First dose of study medication through 6 months after the last dose of study medication

SECONDARY OUTCOMES:
Individual MEDI9090 concentrations | First dose of study medication through 3 months after the last dose of study medication
Number of subjects reporting adverse events | Screening through 3 months after last dose of study medication
Number of subjects reporting serious adverse events | Screening through 3 months after the last dose of study medication
Number of subjects with vital sign abnormalities reported as adverse events | Screening through 3 months after the last dose of study medication
Number of subjects with ECG abnormalities reported as adverse events | Screening through 3 months after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (8):
- United States (5):
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, Huntersville, North Carolina
  - Research Site, San Antonio, Texas
- Japan (3):
  - Research Site, Kōtoku
  - Research Site, Sapporo
  - Research Site, Sunto-gun